CLINICAL TRIAL: NCT03632031
Title: Treatment of Wounds Using Oasis® Extracellular Matrix in the Community Setting
Brief Title: Treatment of Wounds Using Oasis® ECM
Status: Completed | Type: Observational
Sponsor: Cook Biotech Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-001
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Non-healing Wound
Keywords: partial and full-thickness wounds; pressure ulcer; venous ulcer; chronic vascular ulcer; diabetic ulcer
MeSH Terms: conditions — Pressure Ulcer; Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with chronic non-healing wounds: Patients with chronic non-healing wounds with planned use of OASIS Extracellular Wound Matrix
  Interventions: Device: Oasis Extracellular Matrix

INTERVENTIONS:
Device: Oasis Extracellular Matrix — Patients will receive OASIS Extracellular Matrix according to the Instruction for Use

SUMMARY:
The purpose of this clinical study is to gather post-market clinical evidence on the use of Oasis ECM as a treatment for different types of chronic wounds in the community setting in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Non-healing ulcer (any etiology) present for at least 1 month and treated in the ambulatory clinic or home healthcare setting

Exclusion Criteria:

1. Age < 18 years
2. Unable or unwilling to provide informed consent
3. Unable or unwilling to comply with the study follow-up schedule, and procedures
4. Simultaneously participating in another investigational drug or device study
5. Target wound area is < 2 cm2 or > 140 cm2 after baseline debridement
6. Target wound has reduced in area by > 40% with 4 weeks of documented standard of care therapy
7. Known allergy to pig or porcine products
8. Systemic infection
9. Infection of the target wound as determined by the collection of pus
10. Osteomyelitis
11. ABI/TBI < 0.6 obtained within 3 months prior to the screening visit
12. Other exclusions may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-healing ulcer (any etiology) present for at least 1 month and treated in the ambulatory clinic or home healthcare setting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Wound healing | 12 weeks
  To demonstrate the percentage of patients with wounds progressing to at least 50% healing

SECONDARY OUTCOMES:
Wound closure- Percentage | up to 12 weeks
  Percentage of patients with complete wound closure
Wound closure- Mean number of weeks | up to 12 weeks
  mean number of weeks to complete wound closure
Wound closure- Mean Percentage | up to 12 weeks
  Mean percent wound closure
Patient reported Quality of Life measurement | up to 12 weeks
  The Wound Quality of Life (QoL) questionnaire is used for measurement of Health-Related Quality of Life in patients with chronic wounds. The total value of this measurement is derived from an average of 17 questions; each question has a value of a minimum of 1 and a maximum of 5. The lower the score, the better the outcome. Subscales are not combined to compute a total score.
Adverse Events | up to 12 weeks
  Summary of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Atkin, PhD, Principal Investigator — Mid Yorkshire Teaching NHS Trust
Locations (2):
- United Kingdom (2):
  - Nursery Park Health Centre, Ashington
  - Pinderfields Hospital, Wakefield

IPD SHARING:
Plan to Share IPD: No